CLINICAL TRIAL: NCT06992700
Title: Dynamic Perturbation Training for Home-Based Upper Limb Rehabilitation in Chronic Stroke: A Randomized Controlled Trial
Brief Title: Dynamic Perturbation Training for Home-Based Upper Limb Rehabilitation in Chronic Stroke
Acronym: PER ASPERA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, Associate Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER ASPERA
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Stroke; Neurorehabilitation
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic perturbation telerehabilitation (Experimental): Patients in this group will perform the exercises at home with the paretic upper limb wearing the orthosis, © Aurafix, model ORT-07A, characterised by elastic bands that exert resistance on the distal phalanx of the fingers. Patients will be able to request breaks from using the glove and/or interrupt the session at any time. In order to assess adherence, the time of use of the glove by each patient will be quantified over the period of time available.
  Interventions: Device: Dynamic perturbation-based intervention
- Conventional telerehabilitation (Active Comparator): Patients in this group will perform the exercises at home with the paretic upper limb wearing the orthosis (to stabilise the wrist and eliminate this possible confounding variable), but without the springs that determine resistance (i.e., eliminating the elastic resistance that is the subject of this study);
  Interventions: Other: Exercises without dynamic perturbations

INTERVENTIONS:
Device: Dynamic perturbation-based intervention — The patient will be asked to perform simple motor tasks while wearing the glove at home under remote supervision of the staff involved in the study. In this way, in order to complete the task, the patient will be forced to overcome the elastic force and perform the movement with greater control. What is innovative compared to the common application of this device is its purpose: specifically, the orthosis will be used by applying resistance to the distal phalanx of the fingers of the hand characterised by a stenic deficit. Contrary to the usual application, which involves the use of this device to facilitate deficient movements, it is hypothesised that the application of resistance will induce the central nervous system (CNS) to create alternative strategies offering them the variety and difficulty necessary to stimulate adaptation without subjecting them to stress resulting from sudden and excessive levels of challenge.
  Arms: Dynamic perturbation telerehabilitation
Other: Exercises without dynamic perturbations — Patients in this group will perform the exercises at home with the paretic upper limb wearing the orthosis (to stabilise the wrist and eliminate this possible confounding variable), but without the springs that determine resistance (i.e., eliminating the elastic resistance that is the subject of this study);
  Arms: Conventional telerehabilitation

SUMMARY:
Study procedures: After acquiring clinical-demographic, neurophysiological and clinical-functional data to describe the extent of upper limb impairment at baseline at the facilities of the Rehabilitation Medicine Unit (UMR) of the Ferrara University Hospital (Department of Neuroscience), patients will undergo a 10-day home rehabilitation programme (two consecutive weeks, five days a week, two daily sessions of one hour each) with remote supervision by study staff in a randomised manner in two groups:

* Experimental group: patients in this group will perform the exercises at at home with the paretic upper limb wearing the orthosis, © Aurafix, model ORT-07A, characterised by elastic bands that exert resistance on the distal phalanx of the fingers.
* Control group: patients in this group will perform the exercises at home with the paretic upper limb wearing the orthosis (in order to stabilise the wrist and eliminate this potential confounding variable) but without the springs that provide resistance (i.e. eliminating the elastic resistance that is the subject of this study); Assignment to the treatment group will be based on a randomisation list (generated through https://www.random.org/ to obtain a balanced division) established by the Scientific Director of the study and communicated exclusively to the personnel involved in administering the treatment sessions, while it will not be disclosed to the personnel involved in the other phases of the study. This will allow for the division of patients and an evaluation of the effectiveness of the treatment between the two groups to be as objective as possible. At the end of the ten days of treatment, patients will return to the facilities of the UMR of the Ferrara University Hospital and repeat the assessments already carried out at baseline, in order to evaluate pre/post performance differences after the home treatment and the differences between the two groups. Finally, questionnaires will be administered to assess fatigue at the end of each day of treatment and patient satisfaction in relation to this telerehabilitation approach at the end of the ten days. It should be noted that patients allocated to the control group will be offered the opportunity to undergo the same treatment as the experimental group, i.e. using the orthosis, in order to ensure that all participants have an equal opportunity to benefit from the innovative protocol.

Type of subjects to be enrolled: Subjects diagnosed with chronic cerebral stroke (i.e. at least 6 months after the onset of the acute event) among patients attending the UMR of the Ferrara University Hospital on an outpatient/day-hospital basis for current or previous multidisciplinary rehabilitation treatment specific to the needs of the individual patient.

Information/Consent: Each participant will be assessed to determine their preliminary eligibility, informed about the aim and procedures of the study, provided with all necessary information for possible participation in the study and sign the informed consent form.

Suspension procedure: At any time during the trial, participants may suspend or withdraw from the study at their own discretion. Breaks during the sessions are also provided for if the participant experiences fatigue, which is the only expected adverse effect, in line with what generally found in any form of repeated physical exercise. Such suspensions will be granted whenever requested, in order to alleviate the participant's discomfort and promote their full participation in the treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years or older;
* Diagnosis of first cerebral stroke (ischaemic or haemorrhagic) in the chronic phase (i.e. at least 6 months after the onset of the acute event) verified by brain imaging (brain computed tomography and/or magnetic resonance imaging);
* Motor deficit in the upper limb - and in particular in the hand - caused by stroke, not attributable to other conditions or diseases and not such as to preclude the ability to perform movements with the fingers and to perform movements to grasp objects;
* Ability to express informed consent correctly.
* Availability of a webcam and Internet connection at home for remote supervision of activities by the staff involved in the study.

Exclusion Criteria:

* Medical conditions that may interfere with the ability to safely complete the study protocol;
* Cognitive dysfunction that precludes informed consent;
* Severe neuropsychological disorders;
* Severe visual problems;
* Upper limb pain assessed with Visual Analogue Scale (VAS) > 7;
* Severe internal diseases (e.g. cardiopulmonary, renal, hepatic);
* Diseases with inflammatory skin lesions, wounds, sensory and circulatory disorders below the elbow and on the hand in the area of application;
* Contraindications to transcranial magnetic stimulation (TMS) procedures, assessed as indicated by international reference, such as: presence of intracranial metal implants, positive history of epilepsy, frequent migraines, implantable devices (ventricular-peritoneal shunts, pacemakers, intrathecal pumps, intracranial metal implants). It should be noted that the presence of this type of exclusion criterion will preclude the performance of TMS assessments, but not the remaining procedures of the study;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline; End of intervention (after 10 days of two sessions per day)
  An assessment scale designed to quantify upper limb function in patients with brain damage resulting in hemiparesis. It identifies the subject's ability to handle objects of different shapes, sizes, and materials, and is considered an indirect measure of activity limitation. It consists of 19 items in total, and the score ranges from 0 to 57. Higher scores indicate better motor performance.
Jebsen-Taylor Hand Function Test (JTHFT) | Baseline; End of intervention (after 10 days of two sessions per day)
  Standardised and objective assessment test for hand motor function; allows both precision and gross tasks to be assessed during the simulation of everyday tasks. It consists of seven activities (writing, turning a page, lifting small objects and placing them in a container, stacking blocks, simulated feeding, moving an empty container, moving a full container). The total score is calculated based on the time taken for each individual test (shorter times indicate better performance).
Nine Hole Peg Test (9HPT) | Baseline; End of intervention (after 10 days of two sessions per day)
  It assesses finger dexterity in patients with various types of neurological disorders, including stroke, Parkinson's disease, multiple sclerosis, etc. The equipment consists of: a wooden or plastic board with 9 holes (diameter 10 or 15 mm) spaced 32 or 50 mm apart; 9 pegs (diameter 7 mm, length 32 mm); a container for the pegs; a stopwatch. The patient is asked to place each peg in the holes in the board and then remove them and reposition them in the container as quickly as possible. During the test, the time taken to complete the task is calculated, from the moment the first peg is picked up to when the last one is placed back in the container. Alternatively, the number of pegs placed in 50 or 100 seconds is counted. Longer completion times (or fewer pegs moved, depending on the assessment method) indicate poorer performance.
Box and Block Test (BBT) | Baseline; End of intervention (after 10 days of two sessions per day)
  Hand movement dexterity assessment test measures the ability to grasp large objects that do not require fine motor control. It is used with a wide range of patients with neurological disorders, including motor deficits caused by stroke. It consists of a wooden box divided into two halves and 150 wooden cubes placed in the same half. The patient is asked to move as many cubes as possible, one at a time, within 60 seconds. The score is calculated based on the number of cubes the patient manages to transfer. The test is repeated after a period of time to assess the patient's progress. A higher number of cubes indicates better performance.

SECONDARY OUTCOMES:
Resting Motor Threshold | Baseline; End of intervention (after 10 days of two sessions per day)
  Unit of Measure: % of maximum stimulator output Resting Motor Threshold (RMT) will be defined as the minimum stimulation intensity (expressed as a percentage of the maximum stimulator output) required to elicit motor evoked potentials (MEPs) of at least 50 μV in 5 out of 10 consecutive trials from the first dorsal interosseous (FDI) muscle of the paretic limb. Measurements will be performed using a Bistim stimulator (Magstim, UK) with participants at rest. The same stimulation parameters will be applied consistently across sessions.
Modified Ashworth Scale (MAS) | Baseline
  A scale for assessing muscle tone alteration following central nervous system injury in the upper limbs; it is a test of resistance to passive movements of a body segment, and the score ranges from 0 to 4 (the higher the score, the greater the spasticity).
Stroke Impact Scale (SIS) | Baseline; End of intervention (after 10 days of two sessions per day)
  It assesses the types and intensity of support that a person with disabilities may need to best manage relevant activities of daily living. It consists of three sections comprising: i) 49 activities of living, with 49 items, grouped into 6 subscales (activities in the home or community, learning activities throughout life, activities related to employment, health, safety and social activities); ii) an additional scale of legal protection, with 8 items; iii) non-ordinary medical and behavioural support needs divided into two parts with 29 items (medical support needs, behavioural support needs). Sections 1 and 2 require the use of a 5-point Likert scale (0 to 4) that assesses frequency (0 - less than once a month; 4 - every hour or more), daily duration of support (0 - never; 4 - 4 hours or more), and type of support (0 - none; 4 - total physical assistance). A higher number indicates a significant impact of stroke on quality of life.
Numerical Rating Scale for Fatigue (NRS) | At the end of each of the two daily treatment sessions.
  A simple tool for assessing the parameter of 'fatigue'. The patient is asked to quantify the fatigue experienced by indicating the corresponding number on a scale ranging from 0 (no perceived fatigue) to 10 (maximum fatigue imaginable). Higher scores indicate a higher level of perceived fatigue.
Satisfaction questionnaire on the proposed home-based intervention: | End of intervention (after 10 days of two sessions per day)
  Each participant will be asked to complete a satisfaction questionnaire in order to assess the feasibility, tolerability, and satisfaction in relation to the proposed rehabilitation method.
Motor Evoked Potential (MEP) Amplitude | Baseline; End of intervention (after 10 days of two sessions per day)
  Unit of Measure: microvolts (μV) Corticospinal excitability will also be assessed by recording Motor Evoked Potential (MEP) amplitudes from the FDI muscle following 10 single-pulse TMS stimuli delivered over the primary motor cortex (M1) of the affected hemisphere at an intensity of resting motor threshold (RMT) + 20%. Muscle relaxation will be visually confirmed through electromyography (EMG) monitoring before each stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Fadiga, MD PhD, Study Chair — Università degli Studi di Ferrara
Locations (1):
- Ferrara University Hospital, Ferrara, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No